CLINICAL TRIAL: NCT07188012
Title: A Pilot Study for the Safety and Expression of Dystrophin in Skeletal Muscle After SPOT-mRNA03 Administration in Duchenne Muscular Dystrophy (DMD) Patients
Brief Title: Safety and Dystrophin Expression of SPOT-mRNA03 in Duchenne Muscular Dystrophy (DMD) Patients
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai Siponuoyin Biotechnology Co Ltd (Industry)
Collaborators: Shanghai Children's Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FM-T3-SH
Record Dates: First submitted 2025-08-22; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Duchenne Muscular Dystrophy (DMD)
Keywords: Duchenne Muscular Dystrophy; North Star Ambulatory Assessment; Dystrophin; Gene Therapy; Extracellular Vesicles
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — RNA, Messenger

STUDY DESIGN:
Intervention Model Description: 3 patients will receive a low dose and 3 patients will receive a high dose
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Low Dose and High Dose (Other): 3 patients will be administered with low dose and 3 patients will be administered with high dose
  Interventions: Genetic: mRNA

INTERVENTIONS:
Genetic: mRNA — mRNA therapy delivered by extracellular vesicles (EVs)

SUMMARY:
The primary objective of this study is to evaluate the safety and and tolerability of SPOT-mRNA03 administered by intravenous (IV) infusion to DMD patients. In addition, this study will preliminarily investigate the concentration changes in dystrophin mRNA concentration, dystrophin protein expression and engraftment, as well as cytokine profiles and immunogenicity.

DETAILED DESCRIPTION:
This is a FIH, open-label, single-arm, and single-center exploratory clinical study of SPOT-mRNA03 administered via IV infusion for DMD patients. SPOT-mRNA03 is a muscle-targeted extracellular vesicles (EVs) loaded with full-length dystrophin mRNA. The targeting ability of SPOT-mRNA03 is conferred by molecular targeting peptides on the EVs membrane, enabling the delivery of dystrophin mRNA as a gene therapy product for DMD.

The study has two ascending dose cohorts, 5.0 × 10^9 CN dystrophin mRNA / kg and 5.0 × 10^10 CN dystrophin mRNA / kg. The study will have a screening period of 30 days, during which patients or their legal guardian written informed consent will be obtained before screening assessments and eligibility will be determined. A total of 6 eligible subjects will participate in the study with 3 subjects in each dose cohort [No previous treatment with corticosteroids]. All subjects started taking 0.05-0.1mg/kg (adjusted according to the actual clinical situation) tacrolimus or sirolimus orally once daily at D-3 (3 days before initial dose of SPOT-mRNA03) for 4 weeks. All subjects are first administered via intravenous infusion on D1 and then administered twice a week (once every 4 days) for a total of 8 doses.

Four weeks after the initial administration of the subjects in the previous dose cohort, if there are no serious adverse events related to the treatment, it will be determined that the subjects in next dose cohort could be administered after discussion between the investigators and the sponsor. Safety evaluations on subjects are conducted during each administration and follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. According to the requirements of the region/country and/or IRB/IEC, the patient and/or legal guardian have signed a written informed consent form and are aware of all relevant study content.
2. Ambulatory boys aged between 2 to 6 years of age, inclusive who can work without assistance for at least 10 meters.
3. The medical history includes clinical diagnosis of DMD and confirmed Duchenne mutations using validated genetic testing (MLPA and whole genome sequencing).
4. Able to tolerate muscle biopsy under anesthesia and have no contraindications to biopsy.
5. Heart, liver, lung, and kidney functions are sufficient:

   1. The left ventricular ejection fraction (LVEF) should be ≥ 50%;
   2. Forced vital capacity (FVC) > 50% of the expected value, and do not require nighttime ventilation;
   3. Patient's glomerular filtration rate (GFR)>30 mL/min/1.73 m2

Exclusion Criteria:

1. Complications other than DMD that may cause muscle weakness and/or motor dysfunction.
2. There are severe intellectual disabilities (such as severe autism, severe cognitive impairment, and severe behavioral disorders) that, according to the investigator's judgment, can affect the study.
3. Hospitalization for respiratory failure within 8 weeks prior to screening.
4. Asthma or underlying lung diseases that are poorly controlled, such as bronchitis, bronchiectasis, emphysema, or recurrent infectious pneumonia that investigator believes may affect respiratory function.
5. Severe uncontrolled heart failure (NYHA III-IV), including any of the following conditions：

   1. Intravenous administration of diuretics or positive inotropic drugs is required within 8 weeks prior to screening.
   2. Hospitalization due to worsening heart failure or arrhythmia within 8 weeks prior to screening.
6. Abnormal laboratory values considered clinically significant:

   1. GGT > 3 × upper limit of normal
   2. Bilirubin ≥ 3.0 mg/dL
   3. Creatinine ≥ 1.8 mg/dL
   4. Hemoglobin < 8 or > 18 g/dL
   5. White blood cell count > 18,500/μL
7. Arrhythmias that require anti-arrhythmic treatment.
8. Subjects who are undergoing immunosuppressive therapy.
9. Has used other gene therapy, investigational drugs, or any treatment aimed at increasing dystrophin expression.
10. Subjects with a history of major surgeries within 12 weeks prior to the initial infusion or planning to undergo major surgeries (such as scoliosis surgery) during this study.
11. Subjects who are allergic to investigational products or local aesthetic drugs or have a history of severe allergies or genetic allergic reactions.
12. Within 6 months prior to the initial infusion, the subjects are exposed to another investigational drug or have participated in an intervention clinical trial.
13. Subjects with positive hepatitis B core antibody or hepatitis C antibody or HIV antibody during screening.
14. Investigator believes that the presence of any other serious diseases, medical conditions, or chronic drug treatment needs can pose unnecessary risks to gene transfer.

Ages: 2 Years to 6 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Male patients only, as Duchenne muscular dystrophy (DMD) predominantly affects males
Enrollment: 6 (Estimated)
Dates: Start 2025-08-06 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment-Related Adverse Events Following Intravenous (IV) Infusion of SPOT-mRNA03 in DMD patients | From enrollment through 6 months post-treatment
  Safety and tolerability of SPOT-mRNA03 will be assessed by collection and quantification of all adverse events, graded according to Common Terminology Criteria for Adverse Events (CTCAE) v5.0.

SECONDARY OUTCOMES:
Concentration of Dystrophin mRNA in Serum | 16 weeks
  Dystrophin mRNA concentration measured in serum of DMD patients before and after IV infusion of SPOT-mRNA03. Quantification is performed by qPCR.
Concentration of Dystrophin mRNA in Muscles | 4 weeks
  Dystrophin mRNA concentration measured in muscles of DMD patients at baseline and after the last IV infusion (dose 8) of SPOT-mRNA03. Quantification is performed by qPCR.
Percent of Normal Dystrophin Protein Expression in Muscles | 4 weeks
  Dystrophin protein measured in muscles of DMD patients at baseline and after the last IV infusion (dose 8) of SPOT-mRNA03, expressed as percent of the mean wild-type level in healthy individuals without DMD or Becker muscular dystrophy. Quantification is performed by Western Blot.
Percentage of Dystrophin-Positive Fibers in Muscles | 4 weeks
  Fiber intensity and dystrophin-positive fibers measured in muscles of DMD patients at baseline and after the last IV infusion (dose 8) of SPOT-mRNA03. Quantification is performed by Immunohistochemistry (IHC).
Concentration of Cytokines in Serum | 28 weeks
  Immunogenicity assessment will be measured by evaluating the changes of cytokines levels (TNF-α, INF-γ, IL-2, IL-6, and IL-10) in the serum of DMD patients before and after IV infusion of SPOT-mRNA03. Quantification is performed by enzyme-linked immunosorbent assay (ELISA).
Concentration of Anti-Dystrophin Antibody in Serum | 28 weeks
  Anti-dystrophin antibody concentration measured in the serum of DMD patients before and after IV infusion of SPOT-mRNA03. Quantification is performed by enzyme-linked immunosorbent assay (ELISA).

CONTACTS AND LOCATIONS:
Overall Officials: Wang Jiwen, Principal Investigator — Shanghai Children's Medical Center
Locations (1):
- Shanghai Children's Medical Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared as this is an early-phase pilot study

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-03-20): https://cdn.clinicaltrials.gov/large-docs/12/NCT07188012/Prot_SAP_000.pdf